CLINICAL TRIAL: NCT04182087
Title: Cognitive Function Assessment in Patients With Focal Brain Injury
Acronym: LESCOG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Grenoble Institut des Neurosciences (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.036; 2019-A01094-53 (Other: ID RCB)
Record Dates: First submitted 2019-10-04; First posted 2019-12-02 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Focal Brain Injury; Cognition
Keywords: Behavioral performance; Cortical resection; Stroke
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focal Brain Injury: Patients with focal brain injury (post-stroke or post-cortical resection)
  Interventions: Behavioral: Cognitive tasks

INTERVENTIONS:
Behavioral: Cognitive tasks — Attention, language, memory, decision-making or executive functions

SUMMARY:
This research relates to the study of cognitive deficits related to various focal brain lesions and their localizations in the brain.

it involves building a large database of behavioural responses measured during the performance of cognitive tasks in patients with focal brain injury, to allow to better understand function of brain.

DETAILED DESCRIPTION:
The study of patients with focal lesions is at the origin of many key discoveries in the field of neurology and cognitive neuroscience.

There are many mechanisms of injury in the brain. The investigators focus on delineated lesions (as opposed to panencephalic, infectious or traumatic lesions), including stroke, excision of intracranial expansive processes or cortectomies of epileptogenic foci.

At the CHUGA, several hundred patients are hospitalized each year for stroke, several dozen patients are operated on brain tumor and about thirty patients benefit from surgical treatment for their epilepsy.

Post-injury cognitive disorders represent a large heterogeneous class of neurological disorders. They are differentiated by various clinical and neuropsychological profiles involving different higher functions such as attention, language, memory, decision-making or executive functions. This variability observed in these disorders complicates their characterization. Especially, there is no, on a sufficiently large scale, data collection to establish whether cognitive deficits are explained by the relative contribution of the type of test used, the location of the lesion, the nature of the pathology and the post-injury delay. This requires a large cohort of patients.

The objective of this project is precisely to build a structure-function database in patients with focal brain injury (post-stroke or post-cortical resection), with the aim of conducting a transnosographic and longitudinal study of brain functions in these patients. To the knowledge of the investigators, this type of approach has not yet been proposed. Such a project should eventually lead to a better understanding of the nature of the cognitive deficits observed in different types of lesions, and to refine the correlations between structures and functions. This project is in line with the objectives set by the University Hospital Federation NeuroPsyNov, which was labeled in 2015 (Dir P. Kahane, fhu-neuropsynov.chu-grenoble.fr) and aims to encourage transnosographic and translational studies of neurological and psychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18-70 years old
* A single, focal anatomical lesion of a given cerebral territory (post vascular, post surgical resection) documented by MRI
* Intellectual ability and understanding of instructions compatible with the cognitive tasks to be performed

Exclusion Criteria:

* Patient deprived of liberty
* Somatic disorder likely to affect cognitive abilities
* Pregnant or nursing woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (Age between 18 and 70 years) patients with focal brain injury (post-stroke or post-cortical resection)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2030-02-06 (Estimated); Study Completion 2030-02-06 (Estimated)

PRIMARY OUTCOMES:
Behavioral performance during cognitive tasks: Exploratory | Data collection will be done on one or more routine visits at 3, 6, 12 or 24 months post lesion (so a maximum of four two-hour sessions)
  Behavioral performance during cognitive tasks evaluating attention, memory, language, executive functions and decision-making (reaction time, error rate, modeling parameters): Aggregated data depending of patient disorders linked to the localization of brain lesion and susceptible to evolve in the time (next 10 years).

SECONDARY OUTCOMES:
Behavioral performance (reaction time, error rate, modeling parameters): Exploratory | Data collection will be done on one or more routine visits at 3, 6, 12 or 24 months post lesion (so a maximum of four two-hour sessions)
  Behavioral performance (reaction time, error rate, modeling parameters) for a given localization according to the pathology and the delay relative to the initial event (lesion) (3, 6, 12, 24 months).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kahane, MD, PhD, Principal Investigator — University Hospital, Grenoble; Julien Bastin, PhD, Study Chair — Grenoble Institute of Neurosciences
Locations (1):
- University Hospital, Grenoble, Grenoble, France

REFERENCES:
- [Result] Adolphs R. Human Lesion Studies in the 21st Century. Neuron. 2016 Jun 15;90(6):1151-1153. doi: 10.1016/j.neuron.2016.05.014. PMID 27311080
- [Result] Barbey AK, Colom R, Solomon J, Krueger F, Forbes C, Grafman J. An integrative architecture for general intelligence and executive function revealed by lesion mapping. Brain. 2012 Apr;135(Pt 4):1154-64. doi: 10.1093/brain/aws021. Epub 2012 Mar 6. PMID 22396393
- [Result] Clark L, Bechara A, Damasio H, Aitken MR, Sahakian BJ, Robbins TW. Differential effects of insular and ventromedial prefrontal cortex lesions on risky decision-making. Brain. 2008 May;131(Pt 5):1311-22. doi: 10.1093/brain/awn066. Epub 2008 Apr 3. PMID 18390562
- [Result] Deman P, Bhattacharjee M, Tadel F, Job AS, Riviere D, Cointepas Y, Kahane P, David O. IntrAnat Electrodes: A Free Database and Visualization Software for Intracranial Electroencephalographic Data Processed for Case and Group Studies. Front Neuroinform. 2018 Jul 6;12:40. doi: 10.3389/fninf.2018.00040. eCollection 2018. PMID 30034332
- [Result] Dronkers NF, Wilkins DP, Van Valin RD Jr, Redfern BB, Jaeger JJ. Lesion analysis of the brain areas involved in language comprehension. Cognition. 2004 May-Jun;92(1-2):145-77. doi: 10.1016/j.cognition.2003.11.002. PMID 15037129
- [Result] Kos C, van Tol MJ, Marsman JB, Knegtering H, Aleman A. Neural correlates of apathy in patients with neurodegenerative disorders, acquired brain injury, and psychiatric disorders. Neurosci Biobehav Rev. 2016 Oct;69:381-401. doi: 10.1016/j.neubiorev.2016.08.012. Epub 2016 Aug 12. PMID 27527825
- [Result] Muller NG, Knight RT. The functional neuroanatomy of working memory: contributions of human brain lesion studies. Neuroscience. 2006 Apr 28;139(1):51-8. doi: 10.1016/j.neuroscience.2005.09.018. Epub 2005 Dec 15. PMID 16352402
- [Result] Petersen SE, Posner MI. The attention system of the human brain: 20 years after. Annu Rev Neurosci. 2012;35:73-89. doi: 10.1146/annurev-neuro-062111-150525. Epub 2012 Apr 12. PMID 22524787
- [Result] Rorden C, Karnath HO. Using human brain lesions to infer function: a relic from a past era in the fMRI age? Nat Rev Neurosci. 2004 Oct;5(10):813-9. doi: 10.1038/nrn1521. PMID 15378041
- [Result] Sperber C, Karnath HO. On the validity of lesion-behaviour mapping methods. Neuropsychologia. 2018 Jul 1;115:17-24. doi: 10.1016/j.neuropsychologia.2017.07.035. Epub 2017 Aug 3. PMID 28782546